CLINICAL TRIAL: NCT04488744
Title: Modeling Tobacco Smoking by IV Pulsed Nicotine in Smokers
Brief Title: Smoking by IV Pulsed Nicotine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: MS059
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: placebo-controlled, mixed-design with nicotine dose as a between-subject and nicotine delivery rate as a within-subject factor.
Who Masked: Participant, Investigator
Masking Description: Participant will not know nicotine dose or rate of infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- nicotine infusion 0.2mg (Experimental): nicotine infusion
  0.2 mg nicotine delivered over 2.5 minutes (5 pulsed-nicotine deliveries) The day order will be randomized over 5 days.
  Interventions: Drug: Nicotine 0.2mcg/kg/s and 1.0mcg/kg/s
- nicotine infusion 2.0mg (Experimental): 0.2mg nicotine delivered over 10 min (20 pulsed-nicotine deliveries),
  Interventions: Drug: Nicotine 0.2mcg/kg/s and 1.0mcg/kg/s
- nicotine infusion 1.0mg (Experimental): 1.0 mg nicotine delivered over 2.5 minutes (5 pulsed-nicotine deliveries)
  Interventions: Drug: Nicotine 0.2mcg/kg/s and 1.0mcg/kg/s
- nicotine infuison 1.0mg (Experimental): 1.0 mg nicotine delivered over 10 min (20 pulsed-nicotine deliveries).
  Interventions: Drug: Nicotine 0.2mcg/kg/s and 1.0mcg/kg/s
- Saline (Placebo Comparator): saline delivered over 2minutes ,2.5minutes,10 minutes
  Interventions: Drug: Nicotine 0.2mcg/kg/s and 1.0mcg/kg/s

INTERVENTIONS:
Drug: Nicotine 0.2mcg/kg/s and 1.0mcg/kg/s — Nicotine infusion 0.2 mg nicotine delivered over 2.5 minutes (5 pulsed-nicotine deliveries), 0.2mg nicotine delivered over 10 min (20 pulsed-nicotine deliveries), 1.0 mg nicotine delivered over 2.5 minutes (5 pulsed-nicotine deliveries) and 1.0 mg nicotine delivered over 10 min (20 pulsed-nicotine deliveries).
  Other Names: nicotine infusion

SUMMARY:
To establish a dose-effect curve for nicotine's abuse potential as a function of nicotine dose and delivery rate. Pulsed IV nicotine administration will be used as it closely matches nicotine delivery by inhaled tobacco use.

DETAILED DESCRIPTION:
Both sub-studies will enroll male and female tobacco cigarette smokers. This study will examine the feasibility of the proposed study parameters in a total of 10 completers. In a crossover design, participants will be tested under 5 conditions: 0.2 mg nicotine delivered over 2.5 minutes (5 pulsed-nicotine deliveries), 0.2mg nicotine delivered over 10 min (20 pulsed-nicotine deliveries), 1.0 mg nicotine delivered over 2.5 minutes (5 pulsed-nicotine deliveries) and 1.0 mg nicotine delivered over 10 min (20 pulsed-nicotine deliveries). The main outcome measures will be self-report drug effects and urges to smoke cigarettes.

The investigators hypothesize that the abuse potential and alleviation of smoking urges are produced by nicotine as a function of nicotine dose and delivery rate.

This study is complete with 13 enrolled and 10 completers

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 35 years, who have been smoking tobacco cigarettes for at least a year
* smoke ≥ 5 and less than 20 cigarettes per day
* urine cotinine levels > 100 ng/mL consistent with nicotine intake of an active smoker
* not seeking treatment at the time of the study for nicotine dependence
* in good health as verified by medical history, screening examination, and screening laboratory tests; and 6) for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* History of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the subject to be in the study
* regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* current alcohol or substance dependence for any other recreational or prescription drugs other than nicotine
* use of e-cigarettes more than 10 days in the past 30 days
* urine drug screening indicating recent illicit drugs use (with the exception of marijuana)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Heart rate will be used to see the dose effect | During nicotine infusion max of ten minutes
  the dose-effect curves of nicotine dose and delivery rate in heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No